CLINICAL TRIAL: NCT01075347
Title: Clinical Study: Topical Autologous Serum Application for the Treatment of Corneal Epithelium Defect After Ocular Surgeries
Brief Title: Topical Autologous Serum Application for the Treatment of Corneal Epithelium Defect After Ocular Surgeries
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: We-Li Chen , MD, Natinal Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200701021R
Record Dates: First submitted 2008-12-04; First posted 2010-02-25 (Estimated); Results first posted 2010-09-02 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Corneal Epithelial Defect; Diabetic Retinopathy; Penetrating Keratoplasty
Keywords: autoserum; ocular surgery; corneal epithelium healing
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous serum use (Active Comparator): Patients treated with additional 20% autoserum after diabetic vitrectomy or penetrating keratoplasty
  Interventions: Other: autologous serum
- Non-autologous serum use (Placebo Comparator): Patients treated with traditional medication(0.1% betamethasone, 0.3% gentamicin and 0.4% tropicamide eye drops application 4 times daily) after diabetic vitrectomy or penetrating keratoplasty
  Interventions: Other: Non-autologous serum

INTERVENTIONS:
Other: autologous serum — with postoperative 20% autologous serum diluted with preservative-free artificial tear application bi-hourly during waking hours
  Other Names: Autoserum
  Arms: Autologous serum use
Other: Non-autologous serum — without postoperative 20% autologous serum diluted with preservative-free artificial tear application bi-hourly during waking hours
  Arms: Non-autologous serum use

SUMMARY:
Ophthalmology ,cornea Autologous serum has long been known to be effective to promote corneal epithelial wound healing in a variety of ocular surface disorders. However, its effectiveness for corneal epithelial defects due to pars plana vitrectomy (PPV) for diabetic retinopathy and penetrating keratoplasty has seldom been reported. In this study, we plan to perform a prospective study to determine the effectiveness of topical autologous serum as a primary treatment for corneal epithelial defect in patients undergoing vitrectomy for diabetic retinopathy and penetrating keratoplasty. All patients enrolled in this study have received corneal epithelial debridement at the end of the ocular surgeries, namely PPV for diabetic retinopathy and penetrating keratoplasty. The patients were grouped into two treatment groups. In the control group, the patients receive conventional postoperative eye drops including topical steroid, antibiotic and mydriatics. In the experimental group, the patients receive topical autologous serum eye drops in addition to conventional postoperative eye drops. The duration for cornea surface to completely re-epithelize, the incidence of corneal complications due to delayed surface re-epithelization (e.g. infectious corneal ulcer, corneal melting, sterile corneal ulcer, corneal neovascularization), and the incidence of recurrent epithelial break down after initial epithelization will be compared between these two groups. Patients undergoing PPV for diabetic retinopathy and penetrating keratoplasty will be compared separately

DETAILED DESCRIPTION:
Purpose: To evaluate the treatment effect of autologous serum eye drops for promoting corneal epithelium wound healing in patients receiving pars plana vitrectomy (PPV) for diabetic retinopathy and penetrating keratoplasty. Background: During PPV for diabetic retinopathy retinopathy and penetrating keratoplasty, removal of the edematous corneal epithelial layer was usually required in order to obtain a better surgical view or enhance the postoperative epithelial wound healing process. However, delayed epithelial healing was frequently found in these patients after surgeries. In addition, corneal epithelial defect is also frequent found in diabetic patients after PPV even corneal epithelial debridement is not performed during the operation. Autologous serum, the fluid component of full blood after blood clotting, contains a large variety of growth factors, vitamins, and immunoglobulins. These epitheliotropic factors are thought to be responsible for the therapeutic effect of serum observed on ocular surface disorders. The effects of serum to promote epithelial wound healing have been well documented in cell culture system in a variety of epithelial cell types including corneal epithelial cells. Autologous serum eye drops have also been demonstrated to be beneficial in the treatment of persistent corneal epithelial defects. In this study, we planned a prospective study to determine the effectiveness of autologous serum tears as a primary treatment in corneal epithelial defect following vitrectomy in diabetic patients and penetrating keratoplasty.

ELIGIBILITY:
Inclusion Criteria:

* patients with proliferative diabetic retinopathy who's condition need to receive pars plana vitrectomy or patients who need to receive penetrating keratoplasty

Exclusion Criteria:

* For PPV: ocular disease such as limbal stem cell Insufficiency , glaucoma, lagophthalmos
* For penetrating keratoplasty:ocular or systemic disease that would affect epithelial healing, such as severe dry eye, severe lid abnormalities, limbal stem cell deficiency, or corneal anesthesia

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital, department of Ophthalmology
Locations (1):
- National Taiwan University Hospital, department of Ophthalmology, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Chen YM, Hu FR, Huang JY, Shen EP, Tsai TY, Chen WL. The effect of topical autologous serum on graft re-epithelialization after penetrating keratoplasty. Am J Ophthalmol. 2010 Sep;150(3):352-359.e2. doi: 10.1016/j.ajo.2010.03.024. Epub 2010 Jun 25. PMID 20579630

RESULTS

PARTICIPANT FLOW:
Groups:
- Autologous Serum Use: Patients treated with autoserum after diabetic vitrectomy or penetrating keratoplasty
- Non-autologous Serum Use: Patients treated with traditional medication after diabetic vitrectomy or penetrating keratoplasty
Period: Overall Study
Arm/Group | Autologous Serum Use | Non-autologous Serum Use
Started | 82 | 83
Completed | 82 | 83
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autologous Serum Use | Non-autologous Serum Use | Total
Number analyzed (Participants) | 82 | 83 | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 45 | 87
  >=65 years | 40 | 38 | 78
Age Continuous [Mean (Standard Deviation); unit: years] | 60.8 (18.1) | 59.8 (17.6) | 60.3 (19.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 42 | 86
  Male | 38 | 41 | 79
Region of Enrollment [Number; unit: participants]
  Taiwan | 82 | 83 | 165

OUTCOME MEASURES:

1. Primary Outcome: Patients With Corneal Epithelial Healing Time Within 14 Days
Description: Patients were hospitalized and examined daily for graft re-epithelialization, which was the main outcome measure.Corneal epithelial healing(the process which the new corneal epithelial cells regenerated to cover the bare cornea lost of its epithelium, the cornea's outer layer) was recorded daily by slit-lamp examination with fluorescein staining.Patients with post-operative chronic persistent epithelial defects for >14 days after the operation were treated with therapeutic contact lens (TCL) application and followed up as outpatients.
Time Frame: every day till total re-epithelization up to 14 days
Measure: Number; unit: participants
Arm/Group | Autologous Serum Use | Non-autologous Serum Use
Number analyzed (Participants) | 82 | 83
participants | 78 | 73

2. Secondary Outcome: Patients With Corneal Complications Due to Delayed Surface Re-epithelization (e.g. Infectious Corneal Ulcer, Corneal Melting, Sterile Corneal Ulcer, Corneal Neovascularization)
Time Frame: every day till total re-epithelization up to 14 days
Measure: Number; unit: participants
Arm/Group | Autologous Serum Use | Non-autologous Serum Use
Number analyzed (Participants) | 82 | 83
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Autologous Serum Use | Non-autologous Serum Use
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/83
Other Adverse Events (participants affected / at risk) | 0/82 | 0/83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No